CLINICAL TRIAL: NCT01574287
Title: Amino Acid Transport Imaging of Parathyroid Adenomas With Anti-3-[18F]FACBC
Brief Title: Anti-3-[18F]FACBC Imaging of Parathyroid Adenomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David M. Schuster, MD (Other)
Responsible Party: Sponsor-Investigator, David M. Schuster, MD, Sponsor-Investigator, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00051415
Record Dates: First submitted 2012-03-31; First posted 2012-04-10 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Parathyroid Disease
MeSH Terms: conditions — Parathyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FACBC (Experimental)
  Interventions: Drug: FACBC

INTERVENTIONS:
Drug: FACBC — Drug is give intravenously over 2 minutes at time of scan

SUMMARY:
Hyperparathyroidism (excessive production of parathyroid hormone (PTH) usually caused by a small growth called an adenoma in the parathyroid glands) is an increasingly significant medical and public health condition.

Surgery is the only effective management for primary hyperparathyroidism. However; it is sometimes difficult to pinpoint the adenoma, in part because current methods of imaging often fail to identify the parathyroid adenoma in as many as 30% of patients. In reoperative parathyroidectomy for persistent or recurrent hyperparathyroidism, localization plays an even greater role. Unfortunately current multiple imaging methods fail to localize 10-15% these of tumors.

SPECT/CT with the radiotracer 99mTc sestamibi has become the standard method for pinpointing the tumor. This, however, is a challenge because the parathyroid glands usually are located close to the thyroid and the radiotracer 99mTc sestamibi concentrates both in thyroid and parathyroid tissue. Hence there is a need for a tracer/imaging tool that concentrates in the parathyroid but not in the thyroid.

A more sensitive and specific radiotracer/tracking agent would markedly improve the investigators ability to identify parathyroid tumors preoperatively, and thus offer more patients a minimally invasive parathyroidectomy.

anti-3-[18F]FACBC is an amino acid based PET radiotracer which has shown utility in detecting a variety of tumors. In cell culture experiments, anti-3-[18F]FACBC has shown uptake in parathyroid cells greater than thyroid cells. Therefore, the investigators think that this radiotracer may be able to help us identify parathyroid adenomas better than 99mTc sestamibi.

The primary aim of this study is to determine if anti-3-[18F]FACBC PET-CT demonstrates uptake within parathyroid adenomas. 12 patients with a diagnosis of primary hyperparathyroidism will undergo PET-CT using anti-3-[18F]FACBC in addition to the standard 99mTc sestamibi scanning and other imaging as clinically appropriate such as ultrasound, MRI, and/or contrast enhanced CT scanning. Since all these patients undergo surgery routinely, the investigators will then compare findings at surgery to those of the anti-3-[18F]FACBC PET-CT to determine if this radiotracer is worthy of further study in a more comprehensive experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients will have biochemical and/or clinical evidence of primary hyperparathyroidism and be a surgical candidate for definitive parathyroid surgery .
3. Ability to lie still for PET scanning
4. Patients must be able to provide written informed consent

Exclusion Criteria:

1. Age less than 18.
2. Inability to lie still for PET scanning.
3. Cannot provide written informed consent.
4. History of secondary hyperparathyroidism.
5. Positive serum or urine pregnancy test within 24 hours of imaging

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FACBC
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FACBC
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Detection Rate of Parathyroid Adenomas of Anti-3-[18F]FACBC Modality
Description: Detection rate of parathyroid adenomas using anti-3-[18F]FACBC modality is assessed by comparing [18F]FACBC and surgical findings.
Time Frame: At approximately 1 month post scan (time of surgery and pathologic analysis)
Measure: Number; unit: percentage of adenomas detected
Arm/Group | FACBC
Number analyzed (Participants) | 4
percentage of adenomas detected | 80

2. Secondary Outcome: Target-to-background Ratio (TBR) of Anti-3-[18F]FACBC for Blood Pool
Description: To evaluate uptake mechanisms of anti-3-[18F]FACBC, target-to-background ratio (TBR) of anti-3-[18F]FACBC is assessed
Time Frame: 5-10 min after intravenous bolus injection of [18F]fluciclovine
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | FACBC
Number analyzed (Participants) | 4
SUVmax | 1.3 (0.6)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | FACBC
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2013-11-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT01574287/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT01574287/SAP_001.pdf